CLINICAL TRIAL: NCT01811628
Title: Project Impact: A Culturally-Tailored Adherence Intervention for Latino Smokers
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2012-1051; K01CA160670 (NIH)
Record Dates: First submitted 2013-03-11; First posted 2013-03-14 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Tobacco Use Cessation
Keywords: Cancer Prevention; Tobacco Use Cessation; Smokers; Recent quitters; Latino; Hispanic; Information; Interview; Questionnaire; Survey; Audio-recorded
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire + Interview: Latinos and Hispanics who are smokers and recent quitters.
  Interventions: Behavioral: Questionnaire; Behavioral: Interview

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire completion taking about 10-15 minutes.
  Other Names: Survey
Behavioral: Interview — Audio-recorded interview that will last about 1 hour.

SUMMARY:
The goal of this research study is to collect information from Latino and Hispanic smokers and recent quitters about factors that are important to them when they are trying to quit. Researchers want to better understand some of the challenges and problems that Latinos and Hispanics face when they try to quit smoking, and then use that information to design a treatment for future smokers.

DETAILED DESCRIPTION:
If participant decides to take part in this study, they will complete a questionnaire about themselves (such as their age, preferred language, and education level) and their smoking habits. This questionnaire should take about 10-15 minutes to complete.

After participant completes this questionnaire, they will be interviewed by a researcher. During this interview participant will be asked to discuss a variety of topics related to smoking and quitting, such as their experience with attempts to quit smoking and problems they may have had. This interview will last about 1 hour.

The interview will be audio-recorded. Participant's interview answers will later be transcribed (written down) without their name or any other identifying information.

Study participation will be complete after the interview.

This is an investigational study.

Up to 48 people will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age
2. Current smoker (>10 cigarettes per day for the past 3 months) or recently quit Smoking (within the past year) but has not smoked for the past 2 months)
3. Read, understand and speak Spanish
4. Identify as being of Latino (or Hispanic) heritage, ethnicity, or ancestry.

Exclusion Criteria:

1. The self-report of a diagnosis of Schizophrenia, Delusional Disorder, Schizoaffective Disorder or Bipolar Disorder in the past year.
2. The self-report of a diagnosis of a Substance Dependence Disorder other than Nicotine in the past year (i.e., Alcohol Dependence, Amphetamine Dependence, Cannabis Dependence, Cocaine Dependence, Hallucinogen Dependence, Inhalant Dependence, Opioid Dependence, Phencyclidine Dependence, Sedatives, Hypnotics, or Anxiolytic Dependence, or Polysubstance Dependence)
3. Unavailable for a 1.5 hour visit to MD Anderson Cancer Center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants recruited through referrals from community health agencies.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-07-17 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Information Collection From Latino and Hispanic Smokers or Recent Quitters | 1 day
  Primary aim of this study is to conduct in-person qualitative interviews with 48 Latino smokers or recent quitters in order to gather information regarding potential elements to include in a future intervention that will target smoking cessation treatment adherence among Latino smokers. This exploratory and qualitative study will utilize thematic analyses of interview discussions to analyze and derive elements that will ultimately be included in a treatment manual.
  Data analyzed using thematic analysis, enabling recurring themes from the data presented and discussed and opposing cases highlighted. Analyses facilitated by the use of N*Vivo - a software package package specific to qualitative research. A qualitative analyses of the content of the qualitative interviews conducted separately for current smokers and recent quitters.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel A. de Dios, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center website — http://www.mdanderson.org